CLINICAL TRIAL: NCT04307745
Title: Primary Prevention Habits for the Shoulder: Survey of the Sportsman's Entourage
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gofflot Amandine, Phd student, University of Liege
Other Study IDs: 1604
Record Dates: First submitted 2020-03-10; First posted 2020-03-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-11

CONDITIONS: Primary Prevention; Shoulder; Questionnaire and Survey
MeSH Terms: interventions — Primary Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Physiotherapist
  Interventions: Other: Primary prevention
- Doctor
  Interventions: Other: Primary prevention
- Physical trainer
  Interventions: Other: Primary prevention
- Trainer
  Interventions: Other: Primary prevention

INTERVENTIONS:
Other: Primary prevention — The primary prevention that the 4 groups put in place for the upper limp athletes

SUMMARY:
Purpose: To provide an update on the implementation of prevention among overhead athletes by their entourage.

Materiel and method: This study will be conducted by the means of a questionnaire. The target population consisted of doctors, trainers, physical trainer and physiotherapist.

The questionnaire will be validated by experts in each categorie and published on an online survey website

ELIGIBILITY:
Inclusion Criteria:

* Professions: physiotherapist, doctor, trainer or physical trainer

Exclusion Criteria:

* Other professions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population will be physiotherapist, doctor, trainer and physical trainer who are one contact with athletes (upper limb athletes).
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Primary prevention of the shoulder | The questionnaire will last 15 minutes at most

CONTACTS AND LOCATIONS:
Overall Officials: Amandine Gofflot, Principal Investigator — ULiège
Locations (1):
- CHU de Liège, Liège, Belgium